CLINICAL TRIAL: NCT01456507
Title: An Open-Label, Single-Dose, Randomized, Three-Way Crossover Study in Healthy Volunteers to Estimate the Effects of Food and of Sprinkling ALO-02 Pellets on Applesauce on the Bioavailability of Oxycodone and Naltrexone/6- Β -Naltrexol From a Extended Release Pellets-in-Capsule Formulation of Oxycodone 40 Mg With Sequestered Naltrexone 4.8 Mg
Brief Title: Healthy Volunteers Study to Estimate the Effects of Food on the Bioavailability of Oxycodone and Naltrexone/6- Β -Naltrexol From a Extended Release Formulation of Oxycodone With Sequestered Naltrexone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B4531003
Record Dates: First submitted 2011-10-13; First posted 2011-10-20 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: Food effect; bioavailability; oxycodone; sequestered Naltrexone; management of moderate to severe pain
MeSH Terms: interventions — oxycodone naltrexone combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): 1×40 mg ALO-02 capsule administered with 240 mL of water under fasting conditions.
  Interventions: Drug: ALO-02 (Oxycodone Naltrexone)
- B (Experimental): 1×40 mg ALO-02 capsule administered with 240 mL of water under fed conditions (standard high fat breakfast).
  Interventions: Drug: ALO-02 (Oxycodone Naltrexone)
- C (Experimental): 1×40 mg ALO-02 with the ALO-02 pellets sprinkled approximately on one table spoon of applesauce, and administered with 240 mL of water under fasting conditions.
  Interventions: Drug: ALO-02 (Oxycodone Naltrexone)

INTERVENTIONS:
Drug: ALO-02 (Oxycodone Naltrexone) — single dose of ALO-02 capsule under fasting condition
  Arms: A
Drug: ALO-02 (Oxycodone Naltrexone) — single dose of ALO-02 capsule under fed condition
  Arms: B
Drug: ALO-02 (Oxycodone Naltrexone) — ALO-02 with the ALO-02 pellets sprinkled on applesauce, and administered under fasting conditions.
  Arms: C

SUMMARY:
The purpose of this study is to estimate the effects of food and of sprinkling ALO-02 pellets on applesauce on the bioavailability of oxycodone and naltrexone/6- beta-naltrexol from an extended release pellets-in-capsule formulation of oxycodone 40 mg with sequestered naltrexone 4.8 mg.

DETAILED DESCRIPTION:
Bioavailability

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive

Exclusion Criteria:

* Evidence or history of clinically significant diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) to time infinity (inf) of oxycodone | predose, 0.5,1,2,4,6,8,12,14,16,24,36,48 hours post-dose
Area Under the Curve (AUC) to last quantifiable concentration (last) of oxycodone | predose, 0.5,1,2,4,6,8,12,14,16,24,36,48 hours post-dose
Maximum Plasma Concentration (Cmax) of oxycodone | predose, 0.5,1,2,4,6,8,12,14,16,24,36,48 hours post-dose

SECONDARY OUTCOMES:
C24, Tmax (time at maximum concentration) and half-life of oxycodone, as data permit. | predose, 0.5,1,2,4,6,8,12,14,16,24,36,48 hours post-dose
AUClast, AUCinf, and Cmax of naltrexone and 6-beta-naltrexol, as data permit | predose, 1,2,4,8,12,24,48,120 hours post-dose
Adverse events, vital signs, pulse oximetry, and safety laboratory parameters. | over 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4531003